CLINICAL TRIAL: NCT06189547
Title: Master's Student in Gastrointestinal Surgery at the First Affiliated Hospital of Guangzhou Medical University
Brief Title: Impact of 10 Different Prior Cancer History on Survival of Patients Who Underwent Surgery for Second Primary Colorectal Cancer: a Population-based Cohort Study
Status: Completed | Type: Observational
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Gao-Min Chen, Principal Investigator, Guangzhou Medical University
Other Study IDs: GMChen
Record Dates: First submitted 2023-12-09; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Second Primary Colorectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Without prior cancer
- With prior colorectal cancer history
  Interventions: Other: different prior cancer history type
- With prior prostate cancer history
  Interventions: Other: different prior cancer history type
- With prior breast cancer history
  Interventions: Other: different prior cancer history type
- With prior uterine cancer history
  Interventions: Other: different prior cancer history type
- With prior bladder cancer history
  Interventions: Other: different prior cancer history type
- With prior skin cancer history
  Interventions: Other: different prior cancer history type
- With prior lung cancer history
  Interventions: Other: different prior cancer history type
- With prior kidney cancer history
  Interventions: Other: different prior cancer history type
- With prior thyroid cancer history
  Interventions: Other: different prior cancer history type
- With prior stomach cancer history
  Interventions: Other: different prior cancer history type

INTERVENTIONS:
Other: different prior cancer history type — different types of prior cancer history
  Groups: With prior bladder cancer history; With prior breast cancer history; With prior colorectal cancer history; With prior kidney cancer history; With prior lung cancer history; With prior prostate cancer history; With prior skin cancer history; With prior stomach cancer history; With prior thyroid cancer history; With prior uterine cancer history

SUMMARY:
In this study, the investigators collected data with the SEER*Stat software version 8.4.1 (accession number: 20377-Nov2021). The patients with confirmed diagnoses of CRC (site code C18.0-20.9 and C26.0) between 2004 and 2013 were retrieved from the Surveillance, Epidemiology, and End Results (SEER) database. Due to the significant disparity in the number of cancer survivors with various prior cancer types among newly diagnosed CRC patients, the investigators utilized the International Classification of Diseases for Oncology, 3rd edition (ICD-O-3) Site Recode to identify 10 common previous cancer sites, including the colorectum, prostate, breast, uterus, bladder, skin, lung, kidney, thyroid, and stomach. CRC patients with a prior history of cancer originated from one of the 10 sites and surgical CRC patients without a prior history of cancer were enrolled in this study. The exclusion criteria were as follows: (1) Patients with more than one cancer in the past; (2) The patient's age at diagnosis was <18 years old; (3) Patients with incomplete survival data and follow-up information; (4) Patients only had autopsy or death certificate records.

The primary outcomes of this study were overall survival (OS) and cancer-specific survival (CSS). OS was defined as the time from diagnosis to date of death（patients who were still alive at the end of follow-up were considered as censored data. CSS was defined as the time from diagnosis to date of death caused by CRC (patients who deaths from other causes or still alive at the end of follow-up were considered as censored data). The investigators set December 31, 2018, as the cut-off date for follow-up to ensure that all included cases (diagnosed in 2004-2013) were followed for at least 5 years.

Based on prior cancer history, the surgical cases were categorized into two groups: 'Non-prior cancer history' and 'Prior cancer history.' The 'Prior cancer history' group was further subcategorized by the type of prior cancer, including colorectum, prostate, breast, uterus, bladder, skin, lung, kidney, thyroid and stomach. The bias between different Prior cancer history group and Non-prior cancer history group was minimized by Propensity Score Matching (PSM), and the Kaplan-Meier method and log-rank tests were used to compare OS and CSS differences. And then, a multivariate Cox proportional hazards model was performed to estimate the hazard ratios (HR) and 95% confidence interval (CI) to analyze whether different types of prior cancer history impacted the OS and CSS in patients who underwent surgery for spCRC independently. Common demographic and clinicopathological data, including age at diagnosis of spCRC, sex, race, marital status, tumor location of spCRC, pathologic grade of spCRC, TNM stage of spCRC (0-I, II-III, IV and unknown) and chemotherapy status were entered as covariates. Kaplan-Meier curves were also constructed according to the time since first cancer diagnosis (latency), age diagnosed with spCRC, and spCRC stage.

Further analysis was performed to determine the impact of surgery on survival of spCRC patients with different type of prior cancer history. The investigators divided patients into surgical and non-surgical groups based on whether surgery was performed, and then assessed the effect of surgery on survival using the propensity score-adjusted Kaplan-Meier method.

In this study, the baseline characteristics of patients were compared using Chi-square test and Fisher's exact test. A one-to-one propensity score matching (PSM) was performed to reduce the selection bias of the two groups of baseline variables. When performing one-to-one propensity score matching between the prior cancer history group and the non-prior cancer history group, the investigators chose a caliper of 0.2. However, the investigators opted for different calipers when matching the surgical and non-surgical groups because the investigators believe that patients with different prior cancers were in entirely different situations. A two-sided probability value of P ≤ 0.05 was considered statistically significant. R software (version 4.2.3) was used for all statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnoses of CRC (site code C18.0-20.9 and C26.0)
* Diagnosis Year between 2004 and 2013

Exclusion Criteria:

* Patients with more than one cancer in the past
* The patient's age at diagnosis was <18 years old
* Patients with incomplete survival data and follow-up information
* Patients only had autopsy or death certificate records

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We used population-based data from the 9 oldest SEER areas, which represented approximately 9% of the US population.
Sampling Method: Probability Sample
Enrollment: 82770 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
overall survival (OS) | From the initial diagnosis of colorectal cancer, at the end of each month
  OS was defined as the time from diagnosis to date of death（patients who were still alive at the end of follow-up were considered as censored data）.

SECONDARY OUTCOMES:
cancer-specific survival (CSS) | From the initial diagnosis of colorectal cancer, at the end of each month
  CSS was defined as the time from diagnosis to date of death caused by CRC (patients who deaths from other causes or still alive at the end of follow-up were considered as censored data)

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Min Chen, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou H, Huang Y, Qiu Z, Zhao H, Fang W, Yang Y, Zhao Y, Hou X, Ma Y, Hong S, Zhou T, Zhang Y, Zhang L. Impact of prior cancer history on the overall survival of patients newly diagnosed with cancer: A pan-cancer analysis of the SEER database. Int J Cancer. 2018 Oct 1;143(7):1569-1577. doi: 10.1002/ijc.31543. Epub 2018 May 7. PMID 29667174
- [Background] Miller KD, Nogueira L, Devasia T, Mariotto AB, Yabroff KR, Jemal A, Kramer J, Siegel RL. Cancer treatment and survivorship statistics, 2022. CA Cancer J Clin. 2022 Sep;72(5):409-436. doi: 10.3322/caac.21731. Epub 2022 Jun 23. PMID 35736631
- [Background] Bluethmann SM, Mariotto AB, Rowland JH. Anticipating the "Silver Tsunami": Prevalence Trajectories and Comorbidity Burden among Older Cancer Survivors in the United States. Cancer Epidemiol Biomarkers Prev. 2016 Jul;25(7):1029-36. doi: 10.1158/1055-9965.EPI-16-0133. PMID 27371756
- [Background] Murphy CC, Gerber DE, Pruitt SL. Prevalence of Prior Cancer Among Persons Newly Diagnosed With Cancer: An Initial Report From the Surveillance, Epidemiology, and End Results Program. JAMA Oncol. 2018 Jun 1;4(6):832-836. doi: 10.1001/jamaoncol.2017.3605. PMID 29167866
- [Background] Gerber DE, Laccetti AL, Xuan L, Halm EA, Pruitt SL. Impact of prior cancer on eligibility for lung cancer clinical trials. J Natl Cancer Inst. 2014 Sep 24;106(11):dju302. doi: 10.1093/jnci/dju302. Print 2014 Nov. PMID 25253615